CLINICAL TRIAL: NCT06772558
Title: The Potential Mechanism by Which Desflurane Induces Postoperative Cognitive Dysfunction in Elderly Perioperative Patients Involves the Modulation of Cdc42 and Clock Proteins, and Their Related Signaling Pathways.
Brief Title: Desflurane Potentially Induces Postoperative Cognitive Dysfunction in Elderly Patients Undergoing Perioperative Procedures by Modulating Cdc42 and Clock Proteins
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-MER-322
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Avascular Necrosis of the Femoral Head; Coronary Artery Disease (CAD); Benign Prostatic Hyperplasia (BPH); Cholecystitis; Knee Osteoarthritis
MeSH Terms: conditions — Femur Head Necrosis; Coronary Artery Disease; Prostatic Hyperplasia; Cholecystitis; Osteoarthritis, Knee | interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- POCD group (Experimental): Postoperative cognitive dysfunction group
  Interventions: Drug: Desflurane Inhalation; Device: mechanical ventilation (MV)
- Control (Active Comparator): No postoperative cognitive dysfunction group
  Interventions: Drug: Desflurane Inhalation; Device: mechanical ventilation (MV)

INTERVENTIONS:
Drug: Desflurane Inhalation — Anesthesia was maintained with either desflurane, with inhaled concentrations adjusted based on electroencephalogram (EEG) monitoring.
Device: mechanical ventilation (MV) — Following induction, patients underwent mechanical ventilation in volume-controlled (VC) mode. Ventilation parameters were set using a GE Aestiva anesthesia machine (GE Healthcare, Waukesha, Wisconsin, USA): tidal volume 6-8 ml/kg, positive end-expiratory pressure 0 cmH2O, inspiration/expiration ratio 1:2, respiratory rate 16 breaths/min, and inspired oxygen concentration of 41%.

SUMMARY:
This clinical trial investigates whether desflurane induces postoperative cognitive dysfunction (POCD) in elderly patients undergoing perioperative procedures by modulating Cdc42 and Clock proteins. The primary research questions are: (1) Does desflurane administration contribute to POCD in this patient population? and (2) Are alterations in Cdc42 and Clock protein levels associated with desflurane-induced POCD in elderly patients? To address these questions, elderly patients will be administered desflurane for anesthesia maintenance. Postoperative assessments will then compare blood levels of Cdc42 and Clock proteins, and examine related signaling pathways, between a control group and a POCD group.

Study participants will receive desflurane anesthesia maintained at a Bispectral Index (BIS) value of 40-60. Postoperative cognitive function will be assessed on the second day using the Montreal Cognitive Assessment (MoCA), and participants will be categorized into either a control group or a POCD group based on MoCA performance. Cognitive function and blood levels of Cdc42 and Clock proteins will be recorded. Furthermore, the study will also investigate associated signaling pathways.

DETAILED DESCRIPTION:
Study Design:

This study is a prospective, randomized, comparative, non-inferiority clinical trial with blinding of both patients and clinicians. It investigates the non-inferiority of desflurane with respect to its impact on Cdc42 and Clock protein levels following POCD in elderly patients. Patient recruitment was conducted at Baogang Hospital, Inner Mongolia. This study received approval from the Medical Ethics Committee of Baogang Hospital, Inner Mongolia, and was performed in accordance with the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants provided voluntary written informed consent.

Patients:

Sixty patients aged >70 years, with an American Society of Anesthesiologists (ASA) physical status of I-III, undergoing elective surgery requiring desflurane-based general anesthesia between February 2025 and May 2025, were recruited. Participants were randomly assigned to one of two groups (n=30 per group).

Randomization and Blinding:

Block randomization was employed to generate the random allocation sequence, with a block size of six. The random sequence was generated using dedicated software (the blockrand package in R version 4.3.2). Allocation of the sequence was performed by an independent third party, and allocation concealment was achieved using sequentially numbered, sealed, opaque envelopes. The research team was blinded to group allocation throughout the randomization process and was not involved in the generation or allocation of the random sequence.

Intervention:

Anesthesia was administered according to standardized institutional protocols. Patients received 1.5-2 mg/kg propofol, 1-2 mg/kg rocuronium, and 1-2 μg/kg remifentanil for induction. Anesthesia was maintained with either sevoflurane or desflurane, with inhaled concentrations adjusted based on electroencephalogram (EEG) monitoring. Remifentanil was continuously infused at 0.05-0.2 μg/kg/min, with adjustments made to maintain blood pressure and heart rate within ±20% of baseline values. Following induction, patients underwent mechanical ventilation in volume-controlled (VC) mode. Ventilation parameters were set using a GE Aestiva anesthesia machine (GE Healthcare, Waukesha, Wisconsin, USA): tidal volume 6-8 ml/kg, positive end-expiratory pressure 0 cmH2O, inspiration/expiration ratio 1:2, respiratory rate 16 breaths/min, and inspired oxygen concentration of 41%.

Outcomes and Measures:

Postoperative follow-up was conducted in the ward by two specially trained nurses who were blinded to patient allocation. Assessments were performed face-to-face at baseline and on the second postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years
* American Society of Anesthesiologists (ASA) physical status classification I-III
* Scheduled to undergo elective surgery requiring general anesthesia with desflurane
* Able and willing to provide voluntary written informed consent
* Able to understand the study procedures and complete follow-up assessments

Exclusion Criteria:

* Pre-existing diagnosis of dementia or any other neurodegenerative disease that could affect cognitive function
* Preoperative Montreal Cognitive Assessment (MoCA) score < 20
* History of severe psychiatric disorders, including psychosis, severe depression, or bipolar disorder
* Unstable angina, uncontrolled hypertension, or a history of myocardial infarction within the past 6 months
* Severe chronic obstructive pulmonary disease (COPD) with significant respiratory compromise, or other significant respiratory disease
* Severe hepatic or renal impairment, defined as Child-Pugh class C for liver disease, or glomerular filtration rate (GFR) < 30 mL/min/1.73 m2 for kidney disease
* History of stroke, transient ischemic attack (TIA), or other significant neurological disorders
* History of alcohol or drug abuse
* Patients with visual, auditory, or language impairments that would interfere with cognitive testing.
* Known allergy or contraindication to any of the study drugs
* Other conditions at the discretion of the investigator that could interfere with the conduct of the study or the interpretation of the results

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | At baseline (before therapy), at 2 days post-treatment
  MoCA, is a rating system from 0 to 30, where 0 represents "no postoperative cognitive dysfunction" and 30 represents the worst possible postoperative cognitive dysfunction.

SECONDARY OUTCOMES:
Cell division control protein 42 homolog (Cdc42) and Circadian Locomotor Output Cycles Kaput(Clock) | At baseline (before therapy), at 2 days post-treatment
  The normal ranges of Cdc42 and Clock were consistent with preoperative levels. The higher the value, the greater the POCD, and the worse the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026-January 2036
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.